CLINICAL TRIAL: NCT01583114
Title: Preventive Effect of ACE Inhibitor Perindopril)on the Onset or Progression of Left Ventricular Dysfoction in Subjects at a Preclinical Stage From Families With Dilated Cardiomyopathy
Brief Title: PREclinical Mutation CARriers From Families With DIlated Cardiomyopathy and ACE Inhibitors
Acronym: PRECARDIA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: recruitement problem
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C10-44; 2010-023184-18 (EudraCT Number)
Record Dates: First submitted 2012-04-11; First posted 2012-04-23 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Dilated Cardiomyopathy
Keywords: dilated cardiomyopathy; heart failure; genetics; mutation carrier; ACE treatment; preclinical
MeSH Terms: conditions — Cardiomyopathy, Dilated; Heart Failure | interventions — Perindopril

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- perindopril (Experimental)
  Interventions: Drug: perindopril
- placebo (Placebo Comparator): same form, administration, posology, frequency and duration as perindopril
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: perindopril — form:1 tablet contained 5 mg of perindopril; posology: 1 intake per day, initiated at a dose of 2.5 mg (1/2 tablet) per day during one week, then 5 mg (1 tablet) per day during two weeks, then 10 mg (2 tablets), or the maximal dose tolerated, until the end of the study (36 months).
  Other Names: Coversyl
  Arms: perindopril
Drug: placebo — form:1 tablet contained 5 mg placebo; posology: 1 intake per day, initiated at a dose of 2.5 mg (1/2 tablet) per day during one week, then 5 mg (1 tablet) per day during two weeks, then 10 mg (2 tablets), or the maximal dose tolerated, until the end of the study (36 months).
  Arms: placebo

SUMMARY:
This is a multicentre European double-blind,randomized and controlled trial with 2 parallel groups (1 study medication, 1 placebo) in order to analyse the impact of ACE inhibitors (ACEi) in subjects who carry a mutation but have not yet developed DCM (dilated cardiomyopathy).

Objective of the trial: Study the impact of ACE inhibitors (ACEi) in subjects who carry a mutation (leading to a genetic form of heart failure) but have not yet developed DCM.

Context. Dilated Cardiomyopathy (DCM) is one of the leading causes of Heart Failure due to systolic dysfunction and at least 30% of DCM are of familial/genetic origin, usually with autosomal dominant inheritance, and underlying genes and mutations are increasingly identified. Familial Dilated Cardiomyopathy (fDCM) is characterized by age-related penetrance (or delayed-onset), that means that the cardiac expression of the disease (echocardiographic abnormalities) is usually absent for a long period and progressively appears with advanced age, usually after 20 years of age

Hypothesis : ACEi may delay or prevent the occurrence of DCM in these subjects (pre-clinical stage).

Expected results: If the hypothesis is confirmed, and as a consequence, the knowledge derived from basic research (genes identification in DCM) will be translated into clinical practice (early identification of subjects at high risk of developing heart failure through predictive genetic testing) with the development of new therapeutic management (early ACEi) that will help to decrease the morbidity and mortality associated with the disease. This will constitute a paradigm of the development of preventive medicine thanks to the development of genetics in the cardiovascular field.

Subjects who are concerned are ≥18 years of age and ≤60 years, carry a mutation responsible for DCM and are at a preclinical stage of the disease. Total duration of treatment (perindopril versus placebo) is 3 years. A total number of 200 participants will be enrolled (100 in each group) in 7 centres.

DETAILED DESCRIPTION:
This study is part of a broader research program, "INHERITANCE" (INtegrated HEart Research In TrANslational genetics of dilated Cardiomyopathies in Europe) research project, submitted to EU (FP7 European Union, HEALTH-2009-2.4.2-3: Translation of basic knowledge on inherited cardiomyopathies into clinical practice) and accepted in 2009 (Grant agreement n° 241924, global coordinator: Pr Eloisa Arbustini, Pavia, Italy).

* Precardia / clinical trial Principal Investigator: Dr Philippe Charron, Pitié Salpêtrière hospital, France
* FP7 Global Inheritance network coordinator: Pr Eloisa Arbustini, Italia

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 years and ≤60 years
* At least one family member should have a clinical diagnosis of dilated cardiomyopathy (LVEF<45% and LVEDD>112%)and should not be considered as the burn-out phase of another cardiomyopathy (such as HCM, ARVC). LV noncompaction may co-exist with DCM in this patient.NB:in a patient with a mutation in LMNA gene, LVEDD may be normal whereas EF is markedly reduced, so that only a reduced LVEF is mandatory(LVEF<45%).
* Carriers of the mutation that has been identified in the family as associated with DCM, and who have received appropriate genetic counselling before and after the announcement of the genetic result. The mutation within the family should be considered as disease-causing.
* No obvious DCM as assessed by diagnostic criteria indicated elsewhere on echocardiography (WHO & Mestroni et al. 1999 and Mahon et al. 2005: references 3 and 9): LVEF <45% and enlarged LVEDD (>112% of predicted value according to age,BSA).
* Presence of minor LV abnormality:

  * isolated LVEDD > 112% (Henry Formula)
  * or reduced systolic dysfunction: 45% < LVEF < 55%, as assessed on echocardiography.
* Able to provide informed consent, and signed informed consent.
* Able to understand and accept the study constraints
* For some European countries (such as France and Spain): participants (by themselves) should have medical health care coverage to be included in a research study

Exclusion Criteria:

* Other disease or factor that can cause minor LV abnormalities, such as cardiotoxic treatment or significant blood hypertension (with uncontrolled blood pressure or significant hypertrophy on echocardiography).
* Contraindication to ACE inhibitor
* Participants who are already treated with ACE inhibitor, sartan or aldosterone receptor antagonists (for various reason such as arterial hypertension) can not be included in this study, unless they have been off these drugs for a period of 6 weeks before inclusion.
* Impaired renal function: estimated Glomerular Filtration Rate (eGFR), using MDRD formula, < 60 ml/mn/1.73m2.
* Baseline serum potassium >5.5 mmol/L.
* Pregnant, parturient or breastfeeding woman or woman of childbearing potential not under effective contraception or planned pregnancy.
* Participation in another therapeutic trial in the previous 3 months
* Participants treated with lithium
* Participant under legal guardianship

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2011-12; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change in left ventricle diameter / volume / ejection fraction | baseline,12 months, 24 months and 36 months after inclusion
  Primary composite end point:
  * Occurence of DCM (LV ejection fraction LVEF<45% and LVEDD>112%)
  * or deterioration of LV end-diastolic diameter / volume (occurrence of events defined as "+4% LVEDD/LVEDV")
  * or deterioration of Ejection fraction (occurrence of events defined as "-4% LVEF")
  All criteria determined either by Echocardiography (primary end-point 1) or by Magnetic resonance imaging (MRI) primary end-point 2).

SECONDARY OUTCOMES:
Echocardiographic deterioration of LVEDD or Ejection fraction | at baseline and at 24 months and 36 months after inclusion
  Echocardiographic deterioration of LVEDD (comparison of average "final LVEDD compared to baseline LVEDD" between arms) or Ejection fraction (comparison of average "final LVEF vs baseline LVEF" between arms)
MRI - deterioration of LVEDVol or Ejection fraction | at baseline and at 36 months after inclusion
  MRI deterioration of LVEDVol (comparison of average "final LVEDVol compared to baseline LVEDVol" between arms) or Ejection fraction (comparison of average "final LVEF vs baseline LVEF" between arms)
Occurence of DCM (Echo: EF< 45% and LVEDD>112%, ref Mahon, 2005) | baseline, 12 months, 24 months and 36 months after inclusion
  Occurence of DCM on Echocardiography: EF< 45% and LVEDD>112% (ref Mahon, 2005)
Deterioration of other Echocardiographic parameters | at baseline, at 12 months, 24 months and 36 months after inclusion
  Deterioration of other Echocardiographic parameters:
  * TDI velocities (average Sa & Ea velocities) at the mitral annulus (lateral and septal), and the E/Ea ratio
  * strain and strain rate (radial, longitudinal, circonferential strain rate in the basal, mid and apical segments)
  * LV volumes (LVED Vol and LVES Vol, Simpson method, 4 cavity incidence)
Deterioration of hormonal biomarkers in serum | at baseline, at 18 months and 36 months after inclusion
  Deterioration of hormonal biomarkers in serum:
  * Natriuretic peptid: BNP and NTproBNP (+/-4% or final versus baseline).
  * Mid-Regional pro-Adrenomedullin (MR-proADM) and Mid-Regional proANP, (+/-4% or final versus baseline).
Clinical end-point | at each visit (inclusion, at 2 weeks, 3 months, 6 months, then every 6 months to 36 months after inclusion)
  Clinical end-point (statistical power is known to be sufficient):
  * Symptoms: Dyspnoea (NYHA stage 1 to 4)
  * Hospitalisation (not planed) for heart failure
Clinical end-point: death | at each visit (inclusion, at 2 weeks, 3 months, 6 months, then every 6 months to 36 months after inclusion)
  Clinical end-point (statistical power is known to be sufficient):
  * All cause death
  * cardiovascular death (Safety end-point: no excess of)

CONTACTS AND LOCATIONS:
Overall Officials: PHILIPPE CHARRON, Principal Investigator — PITIE SALPETRIERE HOSPITAL, PARIS, FRANCE
Locations (7):
- Skejby University Hospital SUH, Aarhus Universit Hospital, Aarhus, Denmark
- Pitié Salpêtrière Hospital, Paris, France
- University of Heidelberg UKLHD, Heidelberg, Germany
- Academic Hospital IRCCS Foundation Policlinico San Matteo (OSM), Pavia, Italy
- Academisch Medisch Centrum AMC and InterUniversity Institute AMC/ICIN, Amsterdam, Netherlands
- Health in Code SL (SME) - Hospital Marítimo de Oza., A Coruña, Spain
- The Heart Hospital, University College London NHS Foundation Trust, London, United Kingdom